CLINICAL TRIAL: NCT05795556
Title: Biomarkers of Sarcopenia and Frailty in Geriatric Patients
Acronym: BioFrail
Status: Completed | Type: Observational
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Suetta, Professor, MD, Dr.Med., Herlev and Gentofte Hospital
Other Study IDs: H-20057620
Record Dates: First submitted 2023-03-03; First posted 2023-04-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia; Muscle Loss; Fall Patients
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Home-dwelling geriatric outpatients: Home-dwelling geriatric outpatients from the Falls Clinic at Gentofte Hospital .
  Clinical assesment: Blood test, body composition (BIA and/or DXA), balance tests (sway), handgrip strength, isometric knee extension strength, chair-rise test, gait-speed, thickness of the thigh muscles, screening for sarcopenia (SARC-F), screening for malnutrition (SNAQ), screening for depression (GDS-15), screening for self-rated health (EQ-5D-5L), frailty (CSHA Frailty Scale)
  Interventions: Other: Assessing sarcopenia and potential biomarkers of sarcopenia in fall patients

INTERVENTIONS:
Other: Assessing sarcopenia and potential biomarkers of sarcopenia in fall patients — Blood test, body composition (BIA and/or DXA), balance tests (sway), handgrip strength, isometric knee extension strength, chair-rise test, gait-speed, thickness of the thigh muscles (ultrasound), screening for sarcopenia (SARC-F), screening for malnutrition (SNAQ), screening for depression (GDS-15), screening for self-rated health (EQ-5D-5L), frailty (CSHA Frailty Scale)

SUMMARY:
During the last decades there has been an increase in the relative proportion and life expectancy of elderly people. Hence, the number of elderly with diseases and disabilities related to aging will increase and consequently, age-related losses in skeletal muscle mass and physical function represents an important current and future public health issue. Sarcopenia is a progressive and generalized skeletal muscle disorder that is considered central to the development of physical deconditioning and untreated sarcopenia is linked to falls, morbidity, and mortality.

The underlying mechanisms behind the progressive loss of muscle mass and function associated with aging are yet unknown but seems to be multifactorial. A decrease in physical activity level and an altered central and peripheral nervous system innervation have been identified as some of the contributing factors. Furthermore, chronic low-grade inflammation has been proposed as a central contributor to sarcopenia and thus physical frailty.

However, it is not yet clear whether the elevated markers of inflammation seen in the elderly are due to aging, chronic illness, or inactivity. But overall, it seems that inflammation plays an important role in the development of muscle loss, and is related to increased risk of falls, fragility, and early death.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients referred to out-patient clinic for fall assessments
* equal to or over the age of 65

Exclusion Criteria:

* age under 65 years
* participants who do not understand Danish
* severe communicative problems
* moderate to severe dementia or cognitive deficits
* no independent walking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of participants referred to the fall clinic at Gentofte Hospital
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle mass | Baseline
  Determination of skeletal muscle mass measured by Bioelectrical Impedance analysis (BIA Inbody770)
Appendicular lean muscle mass | Baseline
  Determination of appendicular lean muscle mass (The sum of the lean tissue is the arms and legs) measured by Bioelectrical Impedance analysis (BIA Inbody770)
Skeletal muscle mass index (SMI) | Baseline
  Determination of skeletal muscle mass index (The sum of the lean tissue is the arms and legs scaled to height squared (ALM/height(2)) measured by Bioelectrical Impedance analysis (BIA Inbody770)

SECONDARY OUTCOMES:
Muscle Thickness | Baseline
  Determination of muscle thickness of the vastus laterals og rectus femoris assessed by ultrasound
Muscle strength (upper body) | Baseline
  Determination of muscle strength measured by a handgrip dynamometer
Muscle strength (lower body) | Baseline
  Determination of maximal isometric quadriceps muscle strength measured by a handheld dynamometer
Physical Activity (Chair rise) | Baseline
  Determination of physical activity assessed by 30 s sit-to-stand chair rise test and five times sit-to-stand test
Physical Activity (Gait speed) | Baseline
  Determination of physical activity assessed by habitual and maximal 6 meters walking speed
Postural sway | Baseline
  Determination of postural sway will be evaluated with a HUR balance force plate. This device is a precision device that provides objectively measurable data. Thanks to its movable platform, it can measure in all directions. The patients will be performing three balance test; Romberg balance test, tandem test and 15 s one-leg-stand.
SARC-F (sarcopenia screening) | Baseline
  The SARC-F questionnaire is used as a screening tool to identify probable sarcopenia patients. The scores range from 0 to 10, with 0 to 2 points for each component. Studies suggested that a score equal to or greater than 4 is predictive of sarcopenia and poor outcomes.
Geriatric Depression Scale (GDS-15) | Baseline
  GDS-15 is used as a screening tool to facilitate assessment of depression. Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
SNAQ (malnutrition) | Baseline
  The Short Nutritional Assessment Questionnaire (SNAQ) is used as a screening tool to get an insight into patients' nutritional status. Patients with 2 points were classified as moderately malnourished and patients with 3 points or more are classified as severely malnourished.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, Professor, Principal Investigator — Charlotte Suetta
Locations (1):
- Pernille Hansen, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The following will be available: Study Protocol and Statistical Analysis Plan

REFERENCES:
- [Derived] Hansen P, Nygaard H, Praeger-Jahnsen L, Schultz M, Dela F, Aagaard P, Ryg J, Suetta C. GDF-15 plasma levels are elevated in mobility-limited older adults with frailty and sarcopenia-results from the BIOFRAIL study. Geroscience. 2025 Nov 25. doi: 10.1007/s11357-025-01946-6. Online ahead of print. PMID 41286529
- [Derived] Hansen P, Nygaard H, Schultz M, Dela F, Aagaard P, Ryg J, Suetta C. Frailty is associated with a history of falls among mobility-limited older adults-cross-sectional multivariate analysis from the BIOFRAIL study. Eur Geriatr Med. 2025 Aug;16(4):1283-1293. doi: 10.1007/s41999-025-01239-3. Epub 2025 May 27. PMID 40423768
- [Derived] Hansen P, Nygaard H, Ryg J, Kristensen MT, Suetta C. Applying both the 30-s and the 5-repetition sit-to-stand tests captures dissimilar groups and a broader spectrum of physical abilities in mobility-limited older individuals: results from the BIOFRAIL study. Eur Geriatr Med. 2025 Apr;16(2):703-707. doi: 10.1007/s41999-024-01115-6. Epub 2024 Dec 7. PMID 39644455